CLINICAL TRIAL: NCT05360420
Title: Screening and Diagnosis of Nodules ≤2 cm in High-risk HCC Patients in China Based on US and CEUS: a Multicenter, Prospective, Randomized Controlled Study
Brief Title: Diagnosis of Nodules ≤2 cm Based on US and CEUS Compared With Current Clinical Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Third Central Hospital (Other)
Collaborators: Tianjin Second People's Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Peking University Binhai Hospital (Unknown); Tianjin Nankai Hospital (Other); Tianjin Medical University Second Hospital (Other); Tianjin Medical University General Hospital (Other); China-Japan Friendship Hospital (Other); Beijing Hospital (Other Government); Shanxi Province Cancer Hospital (Other); Shanxi Provincial People's Hospital (Other Government); The First Affiliated Hospital of Shanxi Medical University (Other); Second Hospital of Shanxi Medical University (Other); Shengjing Hospital (Other); Hebei General Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); The Third Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: drjingxiang004
Record Dates: First submitted 2022-03-04; First posted 2022-05-04 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Liver Cancer; Liver Cirrhosis
Keywords: Liver Cancer; CEUS; Diagnostic Methods; Cost Optimization
MeSH Terms: conditions — Liver Neoplasms; Liver Cirrhosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate CEUS group (Experimental): CEUS (SonoVue) was performed immediately after routine US screening of suspicious lesions. The lesions were classified according to CEUS examination by the diagnosing physician, including consideration of HCC, suspected HCC, and benign lesions. Further hepatobiliary-specific MRI (Modis/Primexian) was performed for lesions considered HCC or suspicious for HCC, and benign lesions were followed up. The diagnostic findings of hepatobiliary-specific MRI were classified by the diagnosing physician and included consideration of HCC, suspected HCC, and benign lesions. For hepatobiliary-specific MRI lesions considered HCC or suspicious for HCC, pathological examination was performed, and benign lesions were followed up.
  Interventions: Diagnostic Test: Immediate CEUS
- Current clinical procedure group (No Intervention): After the suspicious lesions were screened by routine US, CECT, CEMRI and hepatobiliary-specific MRI (the first enhanced imaging examination) were independently selected by clinicians. According to the first examination results of the contrast-enhanced image, the diagnosis was classified by the diagnosing physician, including considering HCC, suspicious HCC, and benign lesions. Another contrast-enhanced imaging examination (CECT or CEMRI or hepatobiliary-specific MRI or CEUS) was performed again for lesions considered or suspected of HCC (second contrast-enhanced imaging study), and negative lesions were followed up. According to the examination results of the second enhanced imaging, the classification includes considering HCC, suspicious HCC, and benign. Pathological examination was performed for lesions considered HCC or suspicious for HCC on the second enhanced image, and benign lesions were followed up.

INTERVENTIONS:
Diagnostic Test: Immediate CEUS — Subjects will receive CEUS examination immediately for the suspicious lesion detected by US.
  Arms: Immediate CEUS group

SUMMARY:
Due to different etiologies, diagnosis and treatment of HCC in China is different from that in Western countries.US is an important screening method for HCC in patients with liver cirrhosis. CEUS, as an enhanced imaging method based on US, has the advantages of convenience, non-radiation, low cost, short examination time, and the diagnostic performance of HCC is comparable to that of CECT, CEMRI, and hepatobiliary-specific MRI.

It is of great significance to consider the cost-effectiveness of each examination based on the principle of cost minimization. Therefore, we propose immediate CEUS examination for suspicious lesions ≤2 cm screened by US, and determine the diagnostic process of further diagnostic methods based on the CEUS results. The aim of this study is to establish a screening and diagnosis process for HCC ≤2 cm suitable for China considering time effect, economic effect and diagnostic efficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are at high risk of HCC.
2. The ages of patients are between 18 and 80.
3. Patients are with solid liver lesion(s) ≤ 2 cm detected by US.
4. Patient signs the informed consent.

Exclusion Criteria:

1. Patients are with liver cirrhosis due to congenital hepatic fibrosis or due to hepatic vascular diseases such as hereditary telangiectasia, Budd-Chiari syndrome, chronic portal vein occlusion syndrome, congestive heart disease.
2. Patient's age is < 18 years old or > 80 years old.
3. Patients with known hypersensitivity to CEUS, CECT, CEMRI, or hepatobiliary-specific MRI contrast agents.
4. Patient is a pregnant or breastfeeding woman.
5. Patient is not diagnosed based on the reference diagnostic criteria required by the study.
6. Patient is considered to be unsuitable to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6730 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance based on US and immediate CEUS with current routine | 6 to 12 months
  The diagnostic efficacy，including sensitivity, specificity, accurary and AUC， of the two groups for HCC from the detection of suspicious lesions by routine US screening to the final diagnosis.
Time benefits based on US and immediate CEUS with current routine | 6 to 12 months
  Time from the detection of suspicious lesions by routine US screening to the first diagnosis of HCC by enhanced imaging examinations and the final diagnosis of HCC.

SECONDARY OUTCOMES:
The economic benefit based on US and immediate CEUS with current routine | 6 to 12 months
  The cost of imaging studies from the discovery of suspicious lesions by routine US screening to the final clinical diagnosis of HCC or the clinical diagnosis of benign lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Jing, MD, Study Director — Tianjin Third Central Hospital
Locations (1):
- Tianjin Third Central Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No